CLINICAL TRIAL: NCT05953220
Title: Investigating Exposure to Toxicants From Smoking and Vaping in People Using Mental Health Services, a Longitudinal Study
Brief Title: Investigating Exposure to Toxicants From Smoking and Vaping
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS: 314314
Record Dates: First submitted 2023-05-02; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-04

CONDITIONS: Smoking, Tobacco; Vaping; Mental Health Disorder
MeSH Terms: conditions — Tobacco Smoking; Vaping; Mental Disorders | interventions — Smoking Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood samples will be collected at baseline and 6 months for people who smoke, vape or do neither. They be collected at baseline, 3 months and 6 month for people who dual use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Smoking: People who smoke tobacco cigarettes at least daily and have not vaped an e-cigarette (except one or two puffs on a less than monthly basis), used NRT, smoking cessation medication or other tobacco products for the past 6 months.
  Interventions: Other: Exclusive tobacco smoking
- Vaping: People who vape e-cigarettes at least daily and have not smoked tobacco cigarettes (except one or two puffs on a less than monthly basis), used NRT, smoking cessation medication, or any other tobacco product for the past 6 months.
  Interventions: Other: Exclusive e-cigarette use
- Dual: Dual users (predominant vapers): people who vape e-cigarettes at least daily and also smoke cigarettes at least weekly, and have not used NRT, smoking cessation medication, or any other tobacco product for the past 6 months.
  Dual users (predominant smokers): people who smoke tobacco cigarettes at least daily and also vape e-cigarettes at least weekly, and have not used NRT, smoking cessation medication, or any other tobacco product for the past 6 months.
  Interventions: Other: Dual use of e-cigarettes and tobacco smoking
- Non-use: People who have neither smoked, vaped, used NRT, smoking cessation medication, nor any other tobacco product for the past 12 months.
  Interventions: Other: No use of e-cigarettes or tobacco smoking

INTERVENTIONS:
Other: Exclusive tobacco smoking — No intervention, participants own tobacco products
  Groups: Smoking
Other: Exclusive e-cigarette use — No intervention, participants own e-cigarette products
  Groups: Vaping
Other: Dual use of e-cigarettes and tobacco smoking — No intervention, participants own tobacco and e-cigarette products
  Groups: Dual
Other: No use of e-cigarettes or tobacco smoking — No intervention
  Groups: Non-use

SUMMARY:
Background:

Many people who smoke use vaping products to help them quit. Levels of toxicants in urine samples are substantially lower in those who exclusively vape compared to those who smoke, suggesting that vaping poses only a fraction of the harms as smoking. However, vaping is still not risk free, with some studies finding higher levels of some toxicants among vapers compared to those who do not smoke or vape. People with mental health conditions have different smoking patterns compared with the wider general population. It is not known if people with mental health conditions have different vaping pattens, therefore researchers do not know if they are exposed to different levels of vaping related toxicants. Also, smoking exposes people to high levels of polycyclic aromatic hydrocarbons (PAHs), which can reduce the effectiveness of some psychotropic medication and management of symptoms. Vaping exposes people to lower levels of PAHs than smoking, however it is unknown if the levels of PAHs from vaping affect the metabolization of psychotropic medicines.

The goal of this observational study is to learn about levels of tobacco toxicants among people with mental health conditions who vape, smoke, dual use or do neither.

The main question[s] it aims to answer are:

What are the levels of biomarkers of toxicant exposure among those who use community mental health services who exclusively vape, exclusively smoke, dual use or do neither, and how do they change over time? What is the difference in clozapine excretion levels and metabolism among those who use community mental health services who exclusively vape, exclusively smoke or dual use or do neither?

Participants will self report smoking and vaping characteristics and provide blood and urine samples at baseline and six months later. Urine will be analysed for tobacco toxicants. Blood will be analysed for levels of clozapine and other prescribed anti psychotic medication.

Researchers will compare levels of toxicants between people who vape, smoke, dual use, or do neither to see if these is a difference.

DETAILED DESCRIPTION:
This is a longitudinal observational study. It aims to investigate four groups each with 40 participants (160 in total) and follow them up at 6 months (smokers, vapers and non-users) or 3 months and 6 months (dual users). Participants will complete questionnaires and provide urine and blood samples at each data collection session.

Urine samples will be tested for a range of tobacco toxicants and markers of inflammation and oxidative stress. Blood samples will be tested for levels of clozapine an other anti-psychotic medication.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 and over
* People who use community mental health services (including those who attend clozapine clinics)

And one of the 4 categories:

* Exclusive smokers - people who smoke tobacco cigarettes at least daily and have not vaped an e-cigarette (except one or two puffs on a less than monthly basis), used NRT, smoking cessation medication or other tobacco products for the past 6 months.
* Exclusive vapers- people who vape e-cigarettes at least daily and have not smoked tobacco cigarettes (except one or two puffs on a less than monthly basis), used NRT, smoking cessation medication, or any other tobacco product for the past 6 months.
* Dual users- People who smoke tobacco cigarettes at least daily and also vape e-cigarettes at least once a week, and have not used NRT, smoking cessation medication, nor any other tobacco product for the past 6 months.

People who vape e-cigarettes at least daily and also smoke cigarettes at least once a week, and have not used NRT, smoking cessation medication, nor any other tobacco product for the past 6 months.

• Non-users - people who have neither smoked, vaped used NRT, smoking cessation medication, nor any other tobacco product for the past 12 months.

Exclusion Criteria:

* Under the age of 18 years old.
* Unable to give informed consent.
* Unstable mental state defined as 1) severity of symptoms that render the patient unresponsive, unsociable, uncooperative, aggressive 2) memory impairment from head trauma or impaired ability to sustain concentration. To be assessed by clinical recruiting staff from medical records.
* Taking part in another study, experiment or clinical trial in which there is an intervention to alter their smoking/ vaping behaviour.
* Prescribed antibiotics in the past 14 days (recent infection will skew inflammation marker levels)
* Prescribed clozapine less than 18 weeks ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People from London who use community mental health services
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Nicotine | Baseline
  Levels of nicotine and its metabolites (nicotine, 3-hydroxycotinine) in urine
Nicotine | 6 months after baseline
  Levels of nicotine and its metabolites (nicotine, 3-hydroxycotinine) in urine
Tobacco-specific nitrosamines | Baseline
  Levels of NNN, NNK(NNAL), NAB, NAT in urine
Tobacco-specific nitrosamines | 6 months after baseline
  Levels of NNN, NNK(NNAL), NAB, NAT in urine
Volatile organic compounds | Baseline
  Levels of Acrolein, Acrylamide, Acrylonitrile, Benzene and Crotonaldehyde in urine
Volatile organic compounds | 6 months after baseline
  Levels of Acrolein, Acrylamide, Acrylonitrile, Benzene and Crotonaldehyde in urine
Polycyclic aromatic hydrocarbons | Baseline
  Levels of 2-napthol in urine
Polycyclic aromatic hydrocarbons | 6 months after baseline
  Levels of 2-napthol in urine
Metals | Baseline
  Levels of Cadmium, Lead, Mercury, Nickle, Selenium in urine
Metals | 6 months after baseline
  Levels of Cadmium, Lead, Mercury, Nickle, Selenium in urine

SECONDARY OUTCOMES:
Clozapine | Baseline
  Levels of clozapine in blood
Clozapine | 6 months after baseline
  Levels of clozapine in blood

CONTACTS AND LOCATIONS:
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No